CLINICAL TRIAL: NCT05811715
Title: Effects of Whole-body Stretching Exercise During Lunch-break for Reducing Musculoskeletal Pain and Physical Exertion Among Healthcare Professionals
Brief Title: Effects of Whole-body Stretching Exercise for Reducing Musculoskeletal Pain and Physical Exertion Among Healthcare Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 444-37-25613-DS
Record Dates: First submitted 2023-04-01; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthcare Professionals

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): WBS-Whole body stretching exercise group
  Interventions: Other: whole body stretching excercise; Other: educational program
- Group B (Active Comparator): control group
  Interventions: Other: educational program

INTERVENTIONS:
Other: whole body stretching excercise — For the WBS group, each 30 minutes exercise class was run by a one trained physiotherapist to serve a maximum of 10 participants (10 x 3 = 30 participants) working in the hospital. Participants invited to attend the exercise class 3 times a week for 6 weeks in their hospital during lunch-break. During each session, participants asked to perform WBS exercise (Franco et al., 2008).
  Arms: Group A
Other: educational program — Participants received an education program which includes ergonomic principles, WRMSDs and their risk factors, as well as manual handling techniques(Bolbol et al., 2017).

SUMMARY:
Purpose of the study:To investigate effect of whole-body stretching (WBS) exercise during lunch-break for reducing musculoskeletal pain and physical exertion among healthcare professionals

DETAILED DESCRIPTION:
This study involved a single-blinded 2-arm randomized controlled trial (RCT) to compare the effect of WBS exercise versus control group during lunch-break to reduce symptoms of WRMSDs in healthcare professionals. sixty healthcare professionals were recruited from Najran university hospital, Saudi Arabia. Study objectives and procedure were properly explained and written informed consent was obtained at the beginning of the study. All the participants were randomly assigned into two equal groups A and B.

Group A were received the 30 minutes of whole body stretching class while group B were received an education program which includes ergonomic principles, WRMSDs and their risk factors, as well as manual handling techniques were explained .

ELIGIBILITY:
Inclusion Criteria:

* Full time healthcare professionals with more than one year of experience were eligible to participate

Exclusion Criteria:

* Acute musculoskeletal symptoms (pain intensity on visual analogue scale (VAS) > 7)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
musculoskeletal pain | 6 Weeks
  musculoskeletal pain were assessed by Nordic musculoskeletal questionnaire
physical exertion | 6 Weeks
  physical exertion were assessed by Borg rating of perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- Hashim Ahmed, Najrān, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No